CLINICAL TRIAL: NCT04310943
Title: Tislelizumab Combined With Bevacizumab and Albumin Paclitaxel in the Treatment of Advanced Lung Adenocarcinoma: a Single-arm, Phase Ⅱ Clinical Trial
Brief Title: Efficacy and Safety of Tislelizumab Combined With Bevacizumab and Albumin Paclitaxel in Lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Chief Physician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC2003
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Lung Adenocarcinoma Stage IV
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — tislelizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Tislelizumab (200mg,Q3W )+Bevacizumab(15 mg/kg,Q3W)+Albumin paclitaxel(100mg/m2,d1,8,15) for 4 cycles, and if there is no disease progression, patients will receive Tislelizumab(200mg,Q3W) until progression or death.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab, 200mg, Q3W ,use until disease progression
  Other Names: Albumin paclitaxel; Bevacizumab

SUMMARY:
The single arm clinical study is to evaluate the efficacy and safety of Tislelizumab combined with Bevacizumab and albumin paclitaxel in the treatment of advanced lung adenocarcinoma. All of the patients were received EGFR-TKI therapy for 1 line and disease progression. The primary endpoint is six months PFS and safety, the seconday endpoint is ORR and one-year OS rate.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria will receive Tislelizumab combined with Bevacizumab and albumin paclitaxel for 4 cycles. If there is no disease progression, the patient will continue to receive Tislelizumab maintenance therapy, until the disease progresses or death.

ELIGIBILITY:
Inclusion Criteria:

* lung adenocarcinoma stage Ⅳ(according AJCC 8)
* received EGFR-TKI for 1 line and disease progression
* EGFR T790M negative
* ECOG PS 0-2

Exclusion Criteria:

* histology of mixed NSCLC with squamous cell carcinoma, neuroendocrine carcinoma and small cell carcinoma.
* have received checkpoint inhibitor.
* uncontrolled pleural effusion, pericardial effusion, or ascites after appropriate intervention
* any unstable systemic disease
* patients who were treated with systemic glucocorticoids (>10mg/ day prednisone therapeutic dose) or other immunosuppressive drugs within 14 days prior to the initial administration or during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
6m-PFS% | through study completion, an average of 1 year
  The proportion of 6 months progression free survival
Safety of Tislelizumab | 30 days after the trial finished
  TEAE are adverse events that occur during or after the first administration of the study drug until 30 days after the study drug is discontinued or the new anticancer treatment is initiated or worse than at baseline (before treatment)

SECONDARY OUTCOMES:
ORR | one year
  objective response rate
OS rate | one year
  rate of oversurvival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zitvogel L, Galluzzi L, Smyth MJ, Kroemer G. Mechanism of action of conventional and targeted anticancer therapies: reinstating immunosurveillance. Immunity. 2013 Jul 25;39(1):74-88. doi: 10.1016/j.immuni.2013.06.014. PMID 23890065
- [Background] Wallin JJ, Bendell JC, Funke R, Sznol M, Korski K, Jones S, Hernandez G, Mier J, He X, Hodi FS, Denker M, Leveque V, Canamero M, Babitski G, Koeppen H, Ziai J, Sharma N, Gaire F, Chen DS, Waterkamp D, Hegde PS, McDermott DF. Atezolizumab in combination with bevacizumab enhances antigen-specific T-cell migration in metastatic renal cell carcinoma. Nat Commun. 2016 Aug 30;7:12624. doi: 10.1038/ncomms12624. PMID 27571927